CLINICAL TRIAL: NCT02771015
Title: A Mono-centre, Post CE-mark, Prospective-randomized Clinical Trial to Evaluate the Performance of a Flexible Self-adherent Absorbent Dressing Coated With a Soft Silicone Layer After Hip or Knee Arthroplasty or Primary Spine Surgery in Comparison to a Standard Wound Dressing (Cosmopor E®Steril, Fa. Hartmann)
Brief Title: Performance of Flexible Self-adherent Absorbent Dressing Coated With a Soft Silicone Layer After Hip -,Knee- Arthroplasty,Primary Spine Surgery in Comparison to a Standard Wound Dressing
Acronym: wounddressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Jan Bredow, Dr.med., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Uni-Köln_2013-01
Record Dates: First submitted 2015-09-08; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Hip-arthroplasty; Knee-arthroplasty; Spine Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepilex Border® (Active Comparator): Mepilex Border® wound dressing at patients after hip-knee or primary spine surgery
  Interventions: Device: Mepilex Border®
- Cosmopor steril® (Active Comparator): Standard wound dressing at patients after hip-knee or primary spine surgery
  Interventions: Device: Cosmopor steril®

INTERVENTIONS:
Device: Mepilex Border® — randomization
  Arms: Mepilex Border®
Device: Cosmopor steril® — randomization
  Arms: Cosmopor steril®

SUMMARY:
Male or female subjects, 18 years and above, undergoing hip, knee or spinal surgery with an expected hospital stay for 4 days or more will be included in the trial. Individual trial duration will be for 7 days (follow-up). Two hundred subjects will be included in the trial, i.e. 100 subjects per arm. The treatment arm (either new or standard wound dressing) will be assigned by randomization stratified by type of surgery (i.e. hip, knee or spine).

DETAILED DESCRIPTION:
At the baseline visit:

* Subject demographic details
* Inclusion and exclusion criteria
* Vital signs
* Medical and surgical history
* Skin status at incision site
* Mobilisation (subject mobility, mobilisation in bed and chair)
* Medication
* AE/ADE/ SAE/SADE/DD
* Informed consent
* Randomization

At visit 2:

* Type of surgery
* Length of incision
* Intraoperative antibiotic given
* Length of anesthesia

At each visit from visit 3:

* Surgical incision condition (condition under the dressing, condition outside the dressing, exudates amount, exudates nature, wound odour, dressing capacity of handling blood, signs of systemic infection, systemic antibiotic given for the systematic infection, blistering, skin stripping
* Skin status at incision site (type of skin, skin temperature, skin perspiration, oedema, tissue consistency, sensation)
* Mobilisation (subject mobility, mobilisation in bed and chair)
* Dressing change (application and removal)
* Drainage (drainage used, application of the drainage)
* Compression Medication (pain medication and systematic antibiotic treatment)
* Photo (photo before and after dressing removal and if signs of infection)
* Investigator/nurse evaluation (ease of application of the dressing, size of the dressing, shape of the dressing, visibility beneath the dressing, notice any pain at dressing change, ease of removal of the dressing, overall experience)
* Patient evaluation (the patient's overall experience of the dressing, comfort when wearing the dressing).
* Contentious pain - measured by Visual Analog Scale (VAS) Prüfplan: CLOSE 2.0F 28.10.2013 5(40)
* Product application (time application start, time application ended, staff involved, material)
* AE/ADE/SAE/SADE/DD

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18years
2. Have an expected total length of stay of 4 or more days
3. Undergoing elective primary arthroplasty of the hip or knee or spinal surgery
4. Undergoing hip surgery with a standard access
5. Give their written informed consent to participate

Exclusion Criteria:

1. Dressing size does not fit the incision area
2. Known allergy/hypersensitivity to any of the components of the dressing
3. Multi-trauma
4. Undergoing arthroplasty due to tumor
5. Fractures
6. Wound at the surgical site prior to surgery
7. Neurological deficit of operated side (hemiplegia, etc.)
8. Subject has documented skin disease at time of enrolment, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Minimize the Risk of the Development of Blistering | 7 days after surgery
  Number of participants without blisters at study visit

SECONDARY OUTCOMES:
Number of Participants Rated 'Very Good to Excellent' for Comfort, Conformability and the Acceptability of the Dressing | 7 days
  The comfort, conformability and the acceptability of the dressing were measured on all visit in the study, by a study nurses. The patient had to answer questions regarding, the size of the dressing, shape of the dressing, Visibility beneath the dressing, ease of the application of the dressing, ease of removal of the dressing, overall experience of the use of the dressing, notice any pain at dressing change, Comfort of their dressing, overall experience of their dressing. The patient could chose between 1 Good, 2 Very good, 3 Excellent.In most cases, the patient chose very good to excellent for both hip and knee surgery
Comfort, Comformability, Acceptability of the Dressing | 7 days
  The comfort, conformability and the acceptability of the dressing were measured on all visit in the study, by a study nurses. The patient had to answer questions regarding, the size of the dressing, shape of the dressing, Visibility beneath the dressing, ease of the application of the dressing, ease of removal of the dressing, overall experience of the use of the dressing, notice any pain at dressing change, Comfort of their dressing, overall experience of their dressing. The patient could chose between 1 Good, 2 Very good, 3 Excellent
Change From Baseline in Pain on the visual analog scale | 7 days
  Scores range from 0 [no pain] to 10 [worst possible pain]
the overall cost regarding dressing wear time | 7 days
  bill of material costs

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bredow, Principal Investigator — University Hospital Cologne
Locations (1):
- University Hospital Cologne, Cologne, North Rhine-Westphalia, Germany